CLINICAL TRIAL: NCT04516863
Title: Validation of the German Short Version of the Autobiographical Memory Interview in Patients With Depression and Healthy Controls
Brief Title: A Validation Study of the German Autobiographical Memory Interview
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rheinhessen-Fachklinik Alzey (Other)
Collaborators: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Sarah Kayser, PD Dr. med. Sarah Kayser, MSc., Rheinhessen-Fachklinik Alzey
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: D-AMI 1.1
Record Dates: First submitted 2020-08-11; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Retrograde Amnesia
Keywords: Electroconvulsive therapy; Depression; Cognitive side effects
MeSH Terms: conditions — Amnesia, Retrograde; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with depression (Active Comparator): * Major depression according to DSM-V and ICD-10 (ICD F32.1, F32.2, F32.3, F33.1, F33.2, F33.3)
  * Hamilton Depression Rating Scale > 17
  Interventions: Diagnostic Test: German Autobiographical Memory Interview short-form
- Healthy controls (Active Comparator): - Mental health
  Interventions: Diagnostic Test: German Autobiographical Memory Interview short-form

INTERVENTIONS:
Diagnostic Test: German Autobiographical Memory Interview short-form — Diagnostic Test
  Other Names: D-AMI

SUMMARY:
Electroconvulsive therapy (ECT) is recommended for the treatment of severe depression. But, despite the high remission rates the use of ECT is strongly limited by the social stigma and treatment-emergent cognitive side effects in patients. The most relevant is retrograde amnesia (RA), because it can persists for months and years. To measure RA after ECT the short-form of the Autobiographical Memory Interview (SF-AMI) is commonly used. However, the validation of the German SF-AMI has not yet been carried out. Thus, the aim of this study is to validate the German SF-AMI in depressed patient and healthy controls.

The investigators hypothesize that the German SF-AMI is reliable and valid to quantify RA.

DETAILED DESCRIPTION:
To measure retrograde amnesia of autobiographical memory after ECT, various tests were used so far. Currently, the short form of the Autobiographical Memory Interview (AMI-SF) was used most frequently internationally. In Germany there is no validated translation of the AMI-SF. However, in order to be able to systematically record the cognitive side effects of ECT in clinical practice as well as in research in the German-speaking area, it is important to have validated test procedures that can be successfully used in repeated measurements. In this study, the German version of the AMI (D-AMI), i.e. the specificity of the German short version of the autobiographical memory in patients with depression will be investigated. It is also known in healthy people that autobiographical memory contents can no longer be called up over time. Therefore, the aim of this study is to investigate whether a change in autobiographical memory over the course of time in depressed patients differs from healthy control subjects. It should also be shown whether this German short version for examining autobiographical memory (D-AMI) can be carried out.

ELIGIBILITY:
Inclusion Criteria:

* MDD
* HDRS > 17
* Age 18-80
* Ability to give informed consent

Exclusion Criteria:

* Drugs or drug abuse or addictions
* Use of benzodiazepine equivalent to lorazepam> 1.5 mg per day
* Cognitive impairments
* History of traumatic brain injury
* Relevant organic disease, e.g. Multiple sclerosis, Parkinson's disease
* Bipolar illness, dementia or schizophrenic disorder
* German is not the mother tongue
* Inability to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
German Autobiographical Memory Interview short-form | pre-post (six weeks)
  Changes in autobiographical memory measured with the German Autobiographical Memory Interview short-form pre-post in depressed patients vs. a healthy control Group.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HAMD-17) | pre-post (six weeks)
  Change in depression severity
Inventar Depressiver Symptome (IDS) | pre-post (six weeks)
  Change in depression severity
36-item Health Survey (SF-36) | pre-post (six weeks)
  Change in qualtiy of life
Global Self-Evaluation-Memory (GSE-My) | pre-post (six weeks)
  Change in self-evaluation of memory

CONTACTS AND LOCATIONS:
Overall Officials: Sarah PD Dr. med. MSc. Kayser, MD, Principal Investigator — Rheinhessen-Fachklinik Alzey
Locations (1):
- Rheinhessen-Fachklinik Alzey, Alzey, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No